CLINICAL TRIAL: NCT06562166
Title: Online Adaptive Radiotherapy (oART) in Radical Radiotherapy for Cervical Cancer - A Multi-center Randomized Controlled Study
Brief Title: Online Adaptive Radiotherapy for Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The First Affiliated Hospital of Jiangsu University (Unknown); Zhongnan Hospital (Other); Jingzhou First People's Hospital (Unknown); The First Affiliated Hospital of Nanhua University (Unknown); Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ART_cervical cancer
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; adaptive radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ART (Experimental)
  Interventions: Radiation: online adaptive radiotherapy
- IGRT (No Intervention)

INTERVENTIONS:
Radiation: online adaptive radiotherapy — Patients in ART group received daily online adaptive radiotherapy with a prescription dose of 50.4Gy/28f.
  Arms: ART

SUMMARY:
This study aims to evaluate the clinical efficacy and safety of online adaptive radiotherapy for cervical cancer patients received radical radiotherapy. By comparing with image-guided radiotherapy, the study explores the potential advantages of online adaptive radiotherapy in reducing treatment toxicity and improving local control.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. Pathologically confirmed diagnosis of cervical cancer and pathological type of cervical squamous carcinoma;
3. 2018 FIGO Stage Ib3, II, IIIB and IIIC1
4. Proposed radical pelvic radiotherapy + concurrent sensitizing chemotherapy (platinum-based (cisplatin 30-40mg/m2 or carboplatin alone), starting concurrently in the first week, ≥5 courses)
5. ECOG score 0-2
6. Life expectancy greater than 6 months
7. Ability to remain lying down for more than 30 minutes
8. Patients were fully voluntary and autonomous and co-operated in signing the study informed consent form
9. Complete blood count and basal metabolic indexes within 14 days before enrolment must meet the following requirements: NEUT ≥ 1.5*109/L, HGB ≥ 60g/L, platelets ≥ 100×109/, blood creatinine <1.5 mg/dL. AST and ALT are within 2 times the upper limit of normal
10. Must complete baseline assessments and investigations required before treatment before enrolment
11. be eligible for regular follow-up

Exclusion Criteria:

1. Have received radiotherapy or chemotherapy in the past
2. Have undergone radical surgery for cervical cancer
3. Have a previous history of malignant tumor
4. Pregnant or lactating women
5. Presence of other serious co-morbidities such as poorly controlled cardiovascular, urinary, digestive, respiratory, hematological and central nervous system diseases.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Acute non-hematological toxicity | From the start of treatment until 3 months later
  Acute non-hematologic toxicities include gastrointestinal and genitourinary toxicities, which will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
treatment response | 3 months after completion of treatment
  Treatment response will be evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China